CLINICAL TRIAL: NCT06538129
Title: Assessment of Er:YAG Laser for the Control of Hypersensitivity During Tooth Whitening With Hydrogen Peroxide: Protocol for a Split-Mouth Controlled Clinical Trial
Brief Title: Assessment of Er:YAG Laser for the Control of Hypersensitivity During Tooth Whitening With Hydrogen Peroxide
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Er:YAG Laser
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Hypersensitivity; Hypersensitivity, Immediate; Hypersensitivity Response
MeSH Terms: conditions — Hypersensitivity; Hypersensitivity, Immediate | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: Split-mouth
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The participants will receive the hypersensitivity prevention protocol with Er:YAG laser in cervical region (central incisor, lateral incisor and canine).
  Interventions: Procedure: Hypersensitivity prevention protocol with Er:YAG laser
- Control Group (Experimental): The participants will receive the hypersensitivity prevention protocol with neutral sodium fluoride gel for 4 minutes (central incisor, lateral incisor and canine).
  Interventions: Procedure: Hypersensitivity prevention protocol with neutral sodium fluoride gel

INTERVENTIONS:
Procedure: Hypersensitivity prevention protocol with Er:YAG laser — 1.Prophylaxis using airflow system with erythritol, potency 5, water regulator 5; 2.Initial assessment of hypersensitivity using visual analogue scale (VAS); 3.Color assessment (canines, central incisors and lateral incisors) with digital spectrophotometer (Vita Easyshade,); 4.Placement of dental dam followed by photoactivation with Valo cordless curing light 5.Hypersensitivity prevention protocol with Er:YAG laser in cervical region (central incisor, lateral incisor and canine); 6.Application of whitening gel (1 mm in thickness) with 35% hydrogen peroxide on maxillary arch (Clareador Whiteness HP; FGM), left to react for 15 minutes; 7.Removal of whitening gel; 8.Repeat procedures (steps 7 and 8); 9.Assessment of hypersensitivity immediately after hypersensitivity prevention procedure, immediately after bleaching, 48 after bleaching and one week after bleaching; 10.Color assessment with digital immediately after bleaching, 48 after bleaching and one week after bleaching.
  Arms: Experimental Group
Procedure: Hypersensitivity prevention protocol with neutral sodium fluoride gel — 1.Prophylaxis using airflow system with erythritol, potency 5, water regulator 5; 2.Initial assessment of hypersensitivity using the VAS; 3.Color assessment (canines, central incisors and lateral incisors) with digital spectrophotometer (Vita Easyshade); 4.Placement of dental dam followed by photoactivation with Valo cordless; 5.Hypersensitivity prevention protocol with neutral sodium fluoride gel for 4 minutes (central incisor, lateral incisor and canine); 6.Application of whitening gel (1 mm in thickness) with 35% hydrogen peroxide on maxillary arch (Clareador Whiteness HP; FGM), left to react for 15 minutes; 7.Removal of whitening gel; 8.Repeat procedures (steps 7 and 8); 9.Assessment of hypersensitivity immediately after hypersensitivity prevention procedure, immediately after bleaching, 48 after bleaching and one week after bleaching; 10.Color assessment with digital spectrophotometer immediately after bleaching, 48 after bleaching and one week after bleaching.
  Arms: Control Group

SUMMARY:
Introduction: Tooth whitening is an aesthetic procedure with rapid results that improves the self-esteem and self-image of patients. However, one of the side effects is dentinal hypersensitivity. The aim of the study is to assess the effectiveness of Er:YAG laser administered prior to bleaching with 35% hydrogen peroxide hypersensitivity.

Methods: The maxillary arch of participants 18 to 45 years of age will be treated using the split-mouth method. Grupo experimental: Hypersensitivity prevention protocol with Er:YAG laser followed by bleaching with 35% hydrogen peroxide; control group: hypersensitivity prevention protocol with neutral sodium fluoride for four minutes followed by bleaching with 35% hydrogen peroxide. Er:YAG laser (2940 nm) will be used with the following parameters: 0.15 W, 10 mJ, 15 Hz and SP mode (pulse duration: 300 µs), TIP: Cylindrical Quartz 1000/4, using the H14 handpiece (H14 for LightWalker AT; Fotona dd, Ljubljana, Slovenia). Each tooth (central incisor, lateral incisor and canine) will be irradiated twice for 10 s in an unfocused scanning motion in the cervical region at a working distance of 1 cm. The absolute risk and intensity of dentinal hypersensitivity during treatment will be assessed using the visual analogue scale. The change in color will be determined using an intraoral spectrophotometer in contact with the tooth. Assessments will be conducted before and after preventive treatment, immediately after treatment as well as 48 hours and one week after treatment. Different statistical tests will be used, with the significance level set at 5% (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* All anterior teeth present without caries or restorations;
* Absence of cervical lesions, dental pain and hypersensitivity prior to treatment;
* Not having previously undergone any tooth whitening procedure.

Exclusion Criteria:

* Smokers;
* Pregnant or nursing women;
* Individuals with gingivitis or periodontitis, those with enamel cracks detected by the transillumination test;
* Those with enamel defects or stains caused by tetracycline;
* Those with systemic diseases;
* Those taking nonsteroidal anti-inflammatory.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Dental Hypersensitivity | At baseline as well as after the hypersensitivity prevention protocol, immediately after bleaching, 48 hours after bleaching and one week after bleaching.
  The patients will be given a questionnaire with the VAS for the measurement of dental hypersensitivity. The patient will indicate the severity of tooth sensitivity by marking a vertical line along a 10-cm horizontal line with 0 (no sensitivity) printed at one end and 10 (severe sensitivity) at the other end for all teeth that receive treatment.

SECONDARY OUTCOMES:
Color assessment (instrumental method) | Before and immediately after bleaching as well as 48 horas and one week after bleaching.
  A contact intraoral spectrophotometer (Vita Easyshade, Vita-Zanhnfabrik, Bad Säckingen, Germany) will be used following the manufacturer's instructions and the method described by Kim-Pusateri et al. (2009). Readings will be made in the central portion of each tooth (central incisors, lateral incisors and canines of the maxillary arch) on twice consecutively. If identical, the values will be recorded. Otherwise, new readings will be made until identical values are achieved. Only one result will be recorded for each tooth.